CLINICAL TRIAL: NCT02331407
Title: Effect of Robot Rehabilitation Exercise Training on Motor Control After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Orentreich Family Foundation (Unknown); Mailman School of Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD3437
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot arm rehabilitation therapy (Experimental): Arm training using the ReoGo robotic device, 3 times a week for 3 weeks.
  Interventions: Device: Robotic arm therapy

INTERVENTIONS:
Device: Robotic arm therapy — Training with the ReoGo device

SUMMARY:
Stroke is a leading cause of neurological disability worldwide, often causing significant weakening and paresis of the affected arm. National spending on post-stroke rehabilitation is project to expand 20% to 35% through 2010. As a new tool for therapists, robotic stroke therapy devices have the potential to be a cost-effective device aid to physical therapy and enable novel modes of exercise not currently available. While recent studies have shown chronic patients benefit from repetitive practice, it is not clear whether they improved via a reduction in impairment or increased functional compensation because there is a lack of standard treatment and scales to assess rehabilitation efficacy in chronic stroke patients. This study aims to reconcile difference performance measurements in robotic rehabilitation to assess the outcome of robotic rehabilitation training.

ELIGIBILITY:
Inclusion Criteria:

1. Hemiparesis of the upper extremity
2. Diagnosis of a first clinically apparent ischemic stroke at least 6 months prior to study entry
3. Age 18 years or older
4. Ability to sit and be active for an hour on a chair (or wheelchair) without cardiac, respiratory disturbances and/or pain.

Exclusion Criteria:

1. Inability to understand and/or follow instructions
2. Pain in shoulder or arm
3. Other neurological or musculoskeletal target organ disorder
4. Inability to give informed consent personally
5. Previous or current contracture of the upper extremity

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Krakauer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Univeristy, Neurological Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with post-stroke arm paresis were recruited from June 2009 to May 2011
Period: Overall Study
Arm/Group | Robot Arm Rehabilitation Therapy
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot Arm Rehabilitation Therapy
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 59 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Stroke Side [Count of Participants; unit: Participants]
  Right | 2
  Left | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Arm Motor Control From Baseline Measured as Average Squared Mahalanobis Distance
Description: Arm motor control was assessed through analysis of reaching movements to targets. We derive a measure of arm motor control using functional principal components analysis of reaching trajectories (average squared Mahalanobis distance). This is a unitless measure and lower change values reflect improvement in motor control, while a higher change value reflect a worsening in motor control.
Time Frame: From baseline to within 1 week post-therapy
Measure: Number; unit: unitless
Arm/Group | Robot Arm Rehabilitation Therapy
Number analyzed (Participants) | 9
unitless | -16.31

2. Secondary Outcome: Fugl-Meyer (FM) Upper Extremity Motor Assessment
Description: The FM is a measure of impairment that considers movement arm, wrist, hand, and coordination. Each of the 22 items is scored on a three-point ordinal scale for total score between a minimum score of 0 and a maximum score of 66. A higher score indicates a better outcome.
Time Frame: baseline (1 and 3 weeks prior to therapy), within 1 week after therapy, 3 weeks after therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robot Arm Rehabilitation Therapy
Number analyzed (Participants) | 9
score on a scale
  Pretest 1: 3 weeks before baseline | 30.3 (15.8)
  Pretest 2: 1 week before baseline | 32.8 (17.4)
  Posttest 1: 1 week after therapy | 36.0 (14.6)
  Posttest 2: 3 weeks after therapy | 38.3 (15.5)

3. Secondary Outcome: Action Research Arm Test
Description: The ARAT tests hand and arm function and consists of 19 items in 4 domains: grasp, grip, pinch, and gross movement. Each domain contains items arranged into hierarchical order of difficulty such that success at the most difficult item of a specific subclass assumes success for all items lower in the hierarchy of the same class. Each item is scored on a four-point ordinal scale for total score between a minimum score of 0 and a maximum score of 57. A higher score indicates a better outcome.
Time Frame: baseline (1 and 3 weeks prior to therapy), within 1 week after therapy, 3 weeks after therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robot Arm Rehabilitation Therapy
Number analyzed (Participants) | 9
score on a scale
  Pretest 1: 3 weeks before baseline | 19.6 (18.0)
  Pretest 2: 1 week before baseline | 21.3 (17.1)
  Posttest 1: 1 week after therapy | 23.7 (18.6)
  Posttest 2: 3 weeks after therapy | 25.0 (16.7)

ADVERSE EVENTS:
Arm/Group | Robot Arm Rehabilitation Therapy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No